CLINICAL TRIAL: NCT00504933
Title: Double-blind, Randomised, Placebo-controlled, Phase III Study Comparing the Efficacy and Safety of Bilastine 20 mg Once Daily and Cetirizine 10 mg for the Treatment of Seasonal Allergic Rhinitis.
Brief Title: Efficacy Study for the Symptomatic Treatment of Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Faes Farma, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BILA 1704/RAE; 2004-004586-14 (EudraCT Number)
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Rhinitis; Allergic; Seasonal; Hay Fever; Pollen Allergy; Pollinosis; Rhinoconjunctivitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis | interventions — bilastine; Cetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Bilastine
  Interventions: Drug: bilastine
- B (Active Comparator): Cetirizine
  Interventions: Drug: Cetirizine
- C (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: bilastine — 20 mg (encapsulated) tablets QD/14days
  Arms: A
Drug: Cetirizine — 10 mg (encapsulated) tablets. QD/14 days
  Other Names: Zyrtec
  Arms: B
Drug: Placebo — (encapsulated) Tablets QD/14 days
  Arms: C

SUMMARY:
The objective of the study is to evaluate the efficacy and tolerability of Bilastine 20 mg, compared to Cetirizine and placebo for the treatment of seasonal allergic rhinitis.

DETAILED DESCRIPTION:
In this pivotal, multicentre, international, randomized, double-blind, placebo and active-comparator controlled, parallel study, 683 patients with SAR will be enrolled. Patients will be required to be 12-70 years old, have SAR for ≥2 years, a positive skin test, total nasal and non-nasal score (TSS) ≥36 (out of 72) during run-in, and a composite instantaneous nasal symptom score ≥6 (out of 12) the morning before randomization. The primary efficacy endpoint will be the AUC of reflective TSS from baseline to Day 14.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex between 12 and 70 years of age.
* Patients with documented clinical history of SAR, for at least 2 years prior to the study inclusion.
* Positive skin prick test for at least one of the seasonal allergen specific of the geographical area.
* A previous positive Prick test, or a positive IgE Test (RAST) may also be accepted for inclusion, if performed within 12 months prior to the inclusion.

Exclusion Criteria:

* Patients who have non-allergic rhinitis (vasomotor, infectious, drug-induced, etc.).
* Negative skin prick test (as defined in point 6.1.1.).
* Patients with nasal polyps or a significant deviation of the nasal septum as judged by the investigator as well as nasal intervention in the previous 6 months. Any other nasal illness that can interfere with the aim of the study.
* Patients who have acute or chronic sinusitis as judged by the investigator.
* Patients who have received anti-allergy immunotherapy in the previous two years or are still receiving this kind of therapy.
* Patients who are taking or have taken specified medications prior to randomisation in the study and have not complied with the specified washout period

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 683 (Actual)
Dates: Start 2005-05; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Area under curve of total symptoms score (TSS) from basal visit to D14 visit, according to the patient's assessment on reflective symptoms. | 14 days

SECONDARY OUTCOMES:
AUC of TSS from baseline to D14 according to the patient's assessments on instantaneous symptoms. | 14 days
Change from baseline at day 7 and day 14 for the following: Patient-rated (reflective and instantaneous) and Investigator-rated (instantaneous; assessed during study visit) TSS, NSS, NNSS and change for each individual symptom. | 14 days
Overall assessment of discomfort caused by SAR using a visual analogue scale (VAS) on day 7 and day 14 vs. day 0.
Investigator-rated Clinical Global Impression (CGI) - assessment of the therapeutic effect and AEs performed at day 14
Responders Rate: responders will be classified based on their TSS decrease from baseline: no responders (<25%), >25%<50%, >50%<75%, >75% and will be described by treatment group with their percentage

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kuna, Prof. Dr, Principal Investigator — Barlicki University Hospital, Medical University of Lodz (Poland)

REFERENCES:
- [Background] Bousquet J, Ansotegui I, Canonica GW, Zuberbier T, Baena-Cagnani CE, Bachert C, Cruz AA, Gonzalez SN, Kuna P, Morais-Almeida M, Mullol J, Ryan DP, Sanchez-Borges M, Valiente R, Church MK. Establishing the place in therapy of bilastine in the treatment of allergic rhinitis according to ARIA: evidence review. Curr Med Res Opin. 2012 Jan;28(1):131-9. doi: 10.1185/03007995.2011.648263. Epub 2011 Dec 22. PMID 22149770
- [Background] Church MK. Safety and efficacy of bilastine: a new H(1)-antihistamine for the treatment of allergic rhinoconjunctivitis and urticaria. Expert Opin Drug Saf. 2011 Sep;10(5):779-93. doi: 10.1517/14740338.2011.604029. Epub 2011 Aug 11. PMID 21831011
- [Background] Jauregui I, Garcia-Lirio E, Soriano AM, Gamboa PM, Antepara I. An overview of the novel H1-antihistamine bilastine in allergic rhinitis and urticaria. Expert Rev Clin Immunol. 2012 Jan;8(1):33-41. doi: 10.1586/eci.11.87. PMID 22149338
- [Result] Kuna P, Bachert C, Nowacki Z, van Cauwenberge P, Agache I, Fouquert L, Roger A, Sologuren A, Valiente R; Bilastine International Working Group. Efficacy and safety of bilastine 20 mg compared with cetirizine 10 mg and placebo for the symptomatic treatment of seasonal allergic rhinitis: a randomized, double-blind, parallel-group study. Clin Exp Allergy. 2009 Sep;39(9):1338-47. doi: 10.1111/j.1365-2222.2009.03257.x. Epub 2009 May 4. PMID 19438584